# An Analysis of Participation Trends: Observing Patient Engagement in Anorexia Nervosa Clinical Trials

An Informed Consent Form For Power Clinical Trial's Anorexia Nervosa Observational Study

Date: January 5, 2024

Introduction to the Informed Consent Form: An Overview

This summary aims to outline our observational clinical study, accentuating its procedures, potential risks, and benefits for participants. Although your consent is necessary, your participation is entirely voluntary, allowing you to withdraw without any repercussions.

Our study seeks to comprehend the rationale behind anorexia nervosa patients' decisions to join, persist, or cease participation in clinical trials. The main procedures encompass completing questionnaires and follow-up calls, tailored to mitigate potential participant risks.

While direct medical benefits may not be immediate in this observational study, the accumulated data will aid in identifying avenues to enhance clinical trial participation rates, ultimately benefiting individuals coping with anorexia nervosa.

The study's findings will yield invaluable insights into the factors influencing clinical trial participation rates. Our aim is to refine recruitment strategies and augment patient engagement in trials, ultimately leading to improved treatment options and outcomes for anorexia nervosa patients. Nonetheless, participation is voluntary, and declining won't affect your rights.

Thoroughly reviewing the consent form and seeking clarification on any concerns before deciding are crucial steps. Engaging in discussions with family, friends, advisors, and healthcare professionals is recommended for an informed decision.

Participation remains entirely voluntary, with the right to withdraw at any time without facing any consequences.

Understanding Factors Influencing Anorexia Nervosa Clinical Trial Participation

Clinical trials play a pivotal role in advancing anorexia nervosa treatments, yet concerns linger about participant representation. This study aims to investigate the factors influencing patient decisions regarding involvement, discontinuation, or re-engagement in anorexia nervosa clinical trials. Uncovering these factors is vital to enhance the relevance and efficacy of future research endeavors.

Ensuring a comprehensive examination, our focus is on recruiting a diverse demographic. We aim to understand how factors such as age, race, income, and education impact participation decisions. This collected data aims to develop more effective strategies for engaging underrepresented groups in future clinical trials.

Participation in this study is entirely voluntary, granting individuals the freedom to withdraw without repercussions. The study procedures, involving questionnaire completion and follow-up calls, pose minimal risks to participants. Prospective participants are strongly encouraged to review the consent form meticulously and seek clarification for any uncertainties.

Ultimately, this trial aims to deepen our understanding of the factors influencing anorexia nervosa clinical trial participation. Improving participation rates could expedite the development of innovative treatments for this challenging condition.

Investigating Anorexia Nervosa Patients' Involvement in Clinical Trials

Our observational clinical research seeks to comprehend the factors guiding anorexia nervosa patients in their choices regarding clinical trial participation—enrollment, withdrawal, and completion. We aim to recruit potential participants from ongoing or past interventional trials, using electronic medical records for identification purposes.

Upon expressing interest, our team will provide an in-depth consent form detailing the study's objectives and the rights of participants. Data collection will involve biweekly questionnaires focused on demographics, medical background, and the motivations behind trial participation. Additionally, we plan to conduct comprehensive quarterly phone or video interviews to gain deeper insights.

The statistical analysis of the amassed data aims to uncover the various factors shaping patient participation in clinical trials. Sharing our findings through conferences and scholarly publications aims to benefit all stakeholders engaged in clinical trials.

Our goal is to utilize these insights to enhance the structure of future clinical studies for anorexia nervosa patients, improving recruitment strategies and bolstering retention rates.

Participation in this study is entirely voluntary, allowing individuals the freedom to withdraw without any repercussions. Minimal risks involve the completion of questionnaires and follow-up interviews. Any inquiries or concerns can be addressed promptly by our easily accessible research team.

Understanding Risks in Anorexia Nervosa Observational Research

Observational clinical studies in anorexia nervosa don't involve experimental therapies, but participation may pose potential risks. These risks may encompass privacy breaches, emotional distress stemming from the study's subject matter, and potential adverse effects due to trial-related procedures.

Before involvement, it's critical to thoroughly read and understand the informed consent form and discuss any concerns with the research team. The team will provide detailed explanations about potential risks, study advantages, and safety precautions implemented to ensure participants' well-being.

Assessing the Potential Advantages of Anorexia Nervosa Observational Trials

Taking part in observational clinical trials centered on anorexia nervosa provides patients with an opportunity to contribute to medical advancements and potentially

improve future treatment options. Despite the lack of experimental therapies, patients can expect attentive care during the study period.

Before committing to trial participation, patients should meticulously evaluate the possible benefits and risks, considering their unique circumstances and goals. Consulting with healthcare providers and the research team is critical for making a well-informed decision.

## Factors to Consider Before Concluding Your Trial Participation

Recognizing that your engagement in a clinical trial may be concluded without your explicit agreement is vital. Researchers or sponsors could terminate the trial due to reasons like study suspension, funding cessation, or if it's in your best interest.

Furthermore, your participation might halt due to health decline, pregnancy, choosing to withdraw after significant updates or non-compliance with study protocols. Reflecting on these aspects before enrolling in a clinical trial is crucial.

### Anorexia Nervosa Clinical Trials: An Analytical Approach

Participating in anorexia nervosa clinical trials is entirely voluntary, granting individuals the option to withdraw without facing any negative implications.

To gain a comprehensive understanding of <u>anorexia nervosa studies</u> worldwide, clinicaltrials.gov, overseen by the National Institutes of Health (NIH), acts as an extensive database. Users can refine their search based on geographic location and specific medical conditions of interest.

Additionally, Power's reference page furnishes an updated directory of ongoing <u>anorexia</u> <u>nervosa clinical trials</u> currently in the recruitment phase.

# Online Resources for Understanding Clinical Trial Diversity

Several online platforms cater to individuals keen on comprehending the intricacies of clinical trial diversity. Here are a couple of articles that might be of interest:

FOX-RAWLINGS, STEPHANIE R., Laura B. Gottschalk, Lauren A. Doamekpor, and Diana M. Zuckerman. "Diversity in medical device clinical trials: do we know what works for which patients?." The Milbank Quarterly 96, no. 3 (2018): 499-529.

<u>Varma, Tanvee, Camara P. Jones, Carol Oladele, and Jennifer Miller. "Diversity in clinical research: public health and social justice imperatives." Journal of Medical Ethics (2022).</u>

These articles provide valuable insights into the challenges faced in achieving diversity in clinical trials and explore potential solutions.

### Preserving Privacy in Research Endeavors

The preservation of confidentiality regarding the data collected in this research is our primary concern. Although complete confidentiality cannot be guaranteed universally, stringent measures are in place to protect it. Keep in mind that legal obligations may mandate the disclosure of personal information. However, any research publications or presentations will maintain your anonymity by refraining from revealing your name or any personally identifying details.

Several entities, such as accrediting bodies, government regulatory authorities (such as the FDA and OHRP), safety monitors, study sponsors, and authorized representatives, may access your medical information for research, quality assurance, and data analysis purposes.

In exceptional cases, we may require an "Authorization Form" outlining the utilization and sharing of your information for this study. Prior to sharing your information or research samples with Power researchers, other university establishments, or external commercial entities for future research, explicit consent will be sought. Your confidential data will be handled securely and appropriately deleted.

# Confirmation of Informed Consent Agreement

By signing this consent agreement, you confirm your understanding and acceptance of the following terms:

• Thorough understanding and comprehension of this informed consent form, with encouragement to seek alternative perspectives before reaching a decision.

- Satisfactory resolution of all your queries regarding the research project and its methodologies, ensuring you possess the necessary information for study participation.
- Consideration of potential benefits, drawbacks, and alternatives linked to participation in the research.
- Assurance that your voluntary involvement in the research study will not restrict your legal rights.
- Prompt communication of any significant updates that might influence your decision to continue participating in the research study.
- Provision of this consent form, allowing you the opportunity to address any remaining questions.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Validation by the Study Investigator | | |
| As the study investigator, I have made certain to address the patient's inquiries comprehensively, ensuring a thorough understanding of the study. Furthermore, I have reaffirmed that the patient's involvement is voluntary and predicated on informed consent. | | |
| Signature of Researcher Who Received Consent | | |
| Name of Investigator | Signature of Investigator | Date |